CLINICAL TRIAL: NCT01747811
Title: Effects of Bright Light Therapy of Sleep, Cognition, Brain Function, and Neurochemistry in Mild Traumatic Brain Injury
Brief Title: Effects of Bright Light Therapy in Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, William D. Killgore, Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-P-001570/1
Record Dates: First submitted 2012-12-06; First posted 2012-12-12 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Concussion, Mild; Post-Concussion Symptoms; Sleep Problems
Keywords: Mild traumatic brain injury; Concussion; Sleep problems; brain imaging; functional magnetic resonance imaging (FMRI)
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- wavelength-1 bright light (Experimental): 30 minutes daily light exposure for 6 weeks
  Interventions: Device: wavelength-1 bright light
- wavelength-2 bright light (Placebo Comparator): 30 minutes daily light exposure for 6 weeks
  Interventions: Device: wavelength-2 bright light

INTERVENTIONS:
Device: wavelength-1 bright light — 6 weeks of daily light exposure, 30 minutes per morning
  Other Names: Philips goLITE energy light
  Arms: wavelength-1 bright light
Device: wavelength-2 bright light — 6 weeks of daily light exposure, 30 minutes per morning
  Other Names: Philips goLITE energy light
  Arms: wavelength-2 bright light

SUMMARY:
Mild traumatic brain injuries (mTBI) or "concussions" are an increasingly prevalent injury in our society. Patients with post-concussion syndrome have been shown to have deficits on tests of short term memory, divided attention, multi-tasking, information processing speed, and reaction time, as well as alteration in mood and emotional functioning. Many patients have other vague complaints including fatigue, dizziness, irritability, sleep disturbances, and chronic headaches. Furthermore, sleep disruption of one of the most common complaints in patients suffering from traumatic brain injuries, with as many as 40 to 65% of patients with mTBI complaining of insomnia. Sleep problems in these patients are associated with poorer outcome, while resolution of the sleep disturbance is associated with improvement in cognitive functioning.

Despite recent evidence of the correlation between sleep quality and recovery from traumatic brain injury, and the well-established role of sleep in neural plasticity and neurogenesis, there have been virtually no direct studies of the causal effects of sleep on recovery following mTBI. However, it is quite likely that sleep plays a critical role in recovery following brain injury.

A particularly promising non-pharmacologic approach that shows potential in improving/modifying abnormalities of the circadian rhythm and sleep-wake schedule is bright light therapy. For the proposed investigation, we hypothesize that bright light therapy may be helpful in improving the sleep of patients with a recent history of mTBI and may also have other mood elevating effects, both of which should promote positive treatment outcome in these individuals. Bright light therapy may increase the likelihood that they will recover more quickly, benefit more extensively from other forms of therapy, and build emotional and cognitive resilience.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18 and 50.
* Subjects must be right handed.
* The primary language of the subjects must be English.
* Subjects have experienced a "concussion" or mTBI within the preceding 18 months, but no sooner that 4 weeks prior to their screening. The occurrence of a concussion or mTBI must be documented by a medical report or other professional witness documentation.
* If documented, Glasgow Coma Scale in the range of 13-15 following the injury.
* Subjects must have complaints of sleep difficulties that emerged or worsened following the most recent head injury.
* At least half of subjects must have evidence of sleep onset insomnia or delayed sleep phase disorder.

Exclusion Criteria:

* Any other history of neurological illness, current Diagnostic and Statistical Manual (DSM-IV) Axis I disorder, lifetime history of psychotic disorder, or head injury with loss of consciousness > 30 minutes
* Complicating medical conditions that may influence the outcome of neuropsychological assessment or functional imaging (e.g., HIV, brain tumor, etc.)
* Mixed or left-handedness
* Abnormal visual acuity that is not corrected by contact lenses
* Contraindicated conditions noted by the manufacture of the light device such as the use of photosynthesizing medications, history of cataract surgery, and pre-existing eye conditions.
* Metal within the body, claustrophobia, or other contraindications for neuroimaging
* Less than 9th grade education
* Excess current alcohol use (more than 2 instances of intake of 5+ drinks (men) when or 4+ drinks (women) when drinking in the past two months, and/or on average drinking > 2 drinks per day (men); > 1 drinks per day (women) during the past two months
* History of alcoholism or substance use disorder
* Significant use of illicit drugs
* History of marijuana use within the past 6 weeks, use of marijuana before the age of 16, and/or use of > 20 marijuana cigarettes throughout the participant's lifetime.
* Subjects who engage in shift-work, night work, or who have substantially desynchronized work-sleep schedules (i.e., sleeping later than 10:00 a.m. more than once a week) will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Killgore, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Bajaj S, Raikes AC, Razi A, Miller MA, Killgore WD. Blue-Light Therapy Strengthens Resting-State Effective Connectivity within Default-Mode Network after Mild TBI. J Cent Nerv Syst Dis. 2021 May 19;13:11795735211015076. doi: 10.1177/11795735211015076. eCollection 2021. PMID 34104033

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Started | 16 | 16
Completed | 14 | 12
Not Completed | 2 | 4
Not completed — Lack of Efficacy | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.07 (7.50) | 23.46 (8.64) | 23.24 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Performance on Multiple Sleep Latency Test (MSLT)
Description: The MSLT is a objective measure of sleepiness. Participants will take a brief nap 3 times during the 1st and second visit. The period of time between wake and sleep onset will be utilized as an objective measure of sleepiness (in minutes). A mean value will be calculated for the entirety of the pre-treatment napping periods and for the post treatment visits.
Time Frame: Change from baseline performance at 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Number analyzed (Participants) | 14 | 12
minutes
  MSLT_PreTreatment_Sleep Onset Latency (SOL) | 6.67 (3.91) | 7.32 (5.41)
  MSLT_PostTreatment_Sleep Onset Latency (SOL) | 6.73 (5.98) | 7.88 (5.83)

2. Secondary Outcome: Neural Activation During Functional Magnetic Resonance Imaging (fMRI) Executive Function Task
Description: Change from baseline in left prefrontal cortical response during a multi source interference task at six weeks. Methods utilized to assess activity in the left prefrontal cortex/inferior frontal operculum included a regions of interest analysis.
Time Frame: Change from baseline performance at 6 weeks (post-treatment)
Population: A total of 22 participants had useable data, 4 participants were excluded due to movement in the images.
Measure: Mean (Standard Deviation); unit: Percent Signal Change
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Number analyzed (Participants) | 13 | 9
Percent Signal Change | 0.098 (0.106) | -0.025 (0.25)

3. Secondary Outcome: Score on Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index is a self report measure of sleep quality. The overall score takes into account many different facets of sleep, such as sleep quality, sleep latency, sleep duration, sleep disturbances, etc. The scores range from 0-21, and any score that is equal to or greater than 5 is indicative of poor sleep quality.
Time Frame: Change from baseline at 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Number analyzed (Participants) | 14 | 12
units on a scale
  Pittsburgh Sleep Quality Index_Mean_PreTreatment | 6.50 (2.14) | 8.25 (1.60)
  Pittsburgh Sleep Quality Index_Mean_PostTreatment | 4.79 (2.29) | 6.25 (3.19)

4. Secondary Outcome: Actigraphy-measured Sleep Quality
Description: Actigraphy is an objective measure that determines sleep vs. wake. It is a watch with an accelerometer worn on the wrist. Sleep quality is determined by the amount of time in bed divided by the amount of time sleeping (in minutes).
Time Frame: Change from baseline at 6 weeks (post-treatment)
Population: We collected usable actigraphy from 29 participants. The 7 remaining participants had unusable actigraphy data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Number analyzed (Participants) | 14 | 12
minutes | 86.17 (1.60) | 85.70 (5.21)

5. Secondary Outcome: Performance on Neuropsychological Assessment
Description: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a neuropsychological assessment that measures different facets of memory including the following: immediate memory, visuospatial/constructional, language, attention, and delayed memory. This is given to all participants on both pre and post treatment visits. The total range for this scale is 40-160. Lower values represent a worse outcome, and higher values represent an improved outcome.
Time Frame: Change from baseline at 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Number analyzed (Participants) | 14 | 12
units on a scale
  Pre-treatment | 102.71 (9.55) | 101.67 (19.01)
  Post Treatment | 98.50 (9.20) | 95.33 (15.39)

6. Other Pre Specified Outcome: Change From Baseline in Beck Depression Inventory (BDI-II) Scores at 6 Weeks
Description: The Beck Depression Inventory (BDI-II) is a self report scale utilized for measuring the severity of depression. Scores can range from 0-63 (0 meaning minimal depressive symptoms, and 63 being severe depressive symptoms). Participants are given this on baseline and post treatment.
Time Frame: Change from baseline at 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Number analyzed (Participants) | 14 | 12
units on a scale | 4.00 (5.07) | 4.83 (3.88)

ADVERSE EVENTS:
Description: No serious or adverse events occurred during the course of the study.
Arm/Group | Wavelength-1 Bright Light | Wavelength-2 Bright Light
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes